CLINICAL TRIAL: NCT01242072
Title: A Phase I Study of Intravenous (IV) Palifosfamide-tris Administered in Combination With IV Etoposide and IV Carboplatin in Patients With Malignancies for Which Etoposide and Carboplatin Are an Appropriate Choice
Brief Title: Intravenous Palifosfamide-tris in Combination With Etoposide and Carboplatin in Patients With Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM1004
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Malignancy; Cancer; Non Small Cell Lung Cancer; Small Cell Lung Cancer; Testicular Cancer; Thymoma; Ovarian Cancer; Osteosarcoma
Keywords: malignancy; etoposide and carboplatin; non small cell lung cancer; small cell lung cancer; testicular cancer; thymoma; ovarian cancer; osteosarcoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Testicular Neoplasms; Thymoma; Ovarian Neoplasms; Osteosarcoma | interventions — isophosphamide mustard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PaCE (Experimental): Palifosfamide, Carboplatin and Etoposide
  Interventions: Drug: palifosfamide-tris

INTERVENTIONS:
Drug: palifosfamide-tris — Intravenous on days 1, 2 and 3 of each 21-day cycle for up to 4 cycles

SUMMARY:
This an an open-label study to define the safety profile and the maximum tolerated dose and confirm the clinical effective dose of palifosfamide-tris given intravenously in combination with etoposide and carboplatin in a wide range of cancers which etoposide and carboplatin are normally given. Once the maximum dose of palifosfamide-tris is determined,a Phase II study using the 3 agents combined will begin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* Malignancy scheduled to receive etoposide and carboplatin therapy
* Eastern Cooperative Oncology Group (ECOG) performance of 0 or 1
* Adequate bone marrow, liver, renal function and coagulation status
* Informed consent
* Agree to use birth control through 28 days of last treatment dose
* Pregnancy test for women of child-bearing potential
* No available standard therapy

Exclusion Criteria:

* Allergy to the the study treatment drugs
* Unstable current medical condition
* Presence or history of injury to the urinary tract
* Active infection
* Major surgery within 4 weeks prior to treatment
* Minor surgery within 2 weeks prior to treatment
* Current acute steroid therapy or taper
* Currently pregnant or nursing
* Substance abuse or condition that may interfere with participation
* Received other investigational drugs within 30 days
* Within 4 weeks of their last chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Assess the safety profile | 21 Days
  Adverse events, vital signs, physical examination, laboratory data and concomitant medications

SECONDARY OUTCOMES:
Determine the maximum tolerated dose | Up to 21 days
  Each dose level cohort will be 3 subjects. After 3 subjects have received a regimen, there will be a minimum observation period of 1 full cycle (21 days) for each of the 3 subjects before enrollment of the group of subjects at the next dose level.
Assess early signs of efficacy | duration of study
  To assess early signs of efficacy using this investigational combination in this patient population

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Research, Lafayette, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - Washington University, St Louis, Missouri